CLINICAL TRIAL: NCT07396415
Title: The Effect of Telehealth-Supported Breastfeeding Counseling on Breastfeeding Duration, Self-Efficacy, and Postpartum Depressive Symptoms: A Randomized Controlled Trial
Brief Title: Telehealth-Supported Breastfeeding Counseling in Primiparous Mothers
Acronym: TELE-BF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MU-SBF-188-2025
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breastfeeding; Postpartum Depression (PPD); Breastfeeding Self-Efficacy
Keywords: Breastfeeding Counseling; Telehealth; Primiparous Mothers; Postpartum Period; Randomized Controlled Trial
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups: a telehealth-supported breastfeeding counseling group or a routine postpartum care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth-Supported Breastfeeding Counseling (Experimental): Participants assigned to this arm will receive structured breastfeeding counseling delivered via telehealth methods, including scheduled video or telephone-based counseling sessions provided by trained healthcare professionals, in addition to routine postpartum care.
  Interventions: Behavioral: Telehealth-Supported Breastfeeding Counseling
- Routine Postpartum Care (Active Comparator): Participants assigned to this arm will receive routine postpartum care according to standard clinical practice, without additional telehealth-supported breastfeeding counseling.
  Interventions: Other: Routine Postpartum Care

INTERVENTIONS:
Behavioral: Telehealth-Supported Breastfeeding Counseling — Structured breastfeeding counseling delivered via telehealth methods, including scheduled video or telephone-based sessions conducted by trained healthcare professionals. The intervention is provided in addition to routine postpartum care and focuses on breastfeeding techniques, problem-solving, maternal support, and breastfeeding self-efficacy during the postpartum period.
  Arms: Telehealth-Supported Breastfeeding Counseling
Other: Routine Postpartum Care — Participants receive routine postpartum care according to standard clinical practice, without additional telehealth-supported breastfeeding counseling.
  Arms: Routine Postpartum Care

SUMMARY:
Breastfeeding is critical for infant and maternal health; however, many first-time mothers experience difficulties that may lead to early discontinuation of breastfeeding. Telehealth-supported breastfeeding counseling has the potential to provide timely, accessible, and continuous support to mothers during the postpartum period.

This randomized controlled trial aims to evaluate the effect of telehealth-supported breastfeeding counseling on breastfeeding duration, breastfeeding self-efficacy, and postpartum depressive symptoms in primiparous mothers. Participants will be randomly assigned to either a telehealth-supported breastfeeding counseling group or a routine postpartum care group.

The intervention group will receive structured breastfeeding counseling sessions delivered via telecommunication tools in addition to standard care, while the control group will receive routine postpartum care only. Outcomes will be assessed using validated questionnaires and follow-up evaluations during the postpartum period. The findings of this study may contribute to improving breastfeeding support strategies and maternal mental health outcomes.

DETAILED DESCRIPTION:
This study is a single-center, parallel-group, randomized controlled trial designed to investigate the effectiveness of telehealth-supported breastfeeding counseling in primiparous mothers.

Eligible participants will be primiparous women who have delivered a healthy, term, singleton infant and meet the inclusion criteria. After providing informed consent, participants will be randomly assigned in a 1:1 ratio to either the intervention group or the control group.

The intervention group will receive structured breastfeeding counseling delivered through telehealth methods, including scheduled video or telephone-based counseling sessions conducted by trained healthcare professionals, in addition to routine postpartum care. The control group will receive routine postpartum care alone.

Primary outcomes include breastfeeding self-efficacy and postpartum depressive symptoms, assessed using validated measurement tools. Secondary outcomes include breastfeeding duration and exclusive breastfeeding status during follow-up. Data will be collected at predefined time points during the postpartum period.

The study will be conducted in accordance with ethical principles and has received approval from the Marmara University Faculty of Health Sciences Non-Interventional Clinical Research Ethics Committee. The results of this study are expected to provide evidence regarding the role of telehealth-based breastfeeding support in improving maternal and infant health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women aged 18-45 years.
* Mothers who have delivered a healthy, term (≥37 weeks), singleton infant.
* Ability to communicate in Turkish.
* Willingness to participate in the study and provide informed consent.
* Access to a telephone or internet-enabled device for telehealth communication.

Exclusion Criteria:

* Mothers with severe maternal medical or psychiatric conditions that may interfere with breastfeeding.
* Infants with congenital anomalies or conditions affecting feeding.
* Mothers who require neonatal intensive care admission for their infants.
* Mothers who are unable to participate in telehealth follow-up.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2027-01-25 (Estimated); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy | From baseline (early postpartum period) to 1 month postpartum
  Change in breastfeeding self-efficacy measured using a validated breastfeeding self-efficacy scale.
Postpartum Depressive Symptoms | From baseline (early postpartum period) to 1 month postpartum
  Change in postpartum depressive symptoms assessed using the Edinburgh Postnatal Depression Scale (EPDS).

SECONDARY OUTCOMES:
Exclusive Breastfeeding Status | Up to 6 months postpartum
  Proportion of mothers exclusively breastfeeding their infants during the follow-up period.
Breastfeeding Duration | Up to 6 months postpartum
  Duration of breastfeeding measured as the length of time mothers continue any breastfeeding during the postpartum follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fetzer JC. How a graduate school education can meet the needs of industrial employment. Anal Bioanal Chem. 2002 Jul;373(4-5):209-10. doi: 10.1007/s00216-002-1334-7. No abstract available. PMID 12171026
- [Result] White RA, Thames HD Jr. State vector models of the cell cycle II: The first three moments of the transit time distribution. J Theor Biol. 1979 Mar 7;77(1):141-60. doi: 10.1016/0022-5193(79)90144-9. No abstract available. PMID 449366